CLINICAL TRIAL: NCT04486443
Title: Effect of Music on Pain in Cancer Patients in Palliative Care Service: a Randomized Controlled Study
Acronym: nursingcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: gönül düzgün (Other)
Responsible Party: Sponsor-Investigator, gönül düzgün, IzmrTinaztepeU, Izmir Tinaztepe University
Organization: Izmir Tinaztepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: izmirtinaztepeuni
Record Dates: First submitted 2020-07-14; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Nursing Caries; Pain; Music Therapy
MeSH Terms: conditions — Pain | interventions — Music Therapy; Complementary Therapies

STUDY DESIGN:
Intervention Model Description: Participants individually randomised to one of two "parallel" groups (Özdemir O 2009). It was considered sufficient to select the participants in the intervention and control groups with the similar 3-4 variables including age and gender (Büyüköztürk Ş 2016). Therefore, patients in the intervention and control groups were randomized according to age, gender and disease stage. The coin tossing method was used to determine which group the patients would involve in. All patients continued to use all medications prescribed before, during and after the research, and no interventions and changes were performed to the patients in this regard. Pain scores of all patients were at 3 and above and they received narcotic analgesics. Researcher generated the allocation sequence, enrolled participants, and assigned participants to interventions.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group received music therapy in 10-minutes sessions with the support of a specialist using the Turkish classical music (Hejaz and Rast modes) accompanied by a tambour. All forms were applied to the group before the music therapy, respectively. Prior to musical therapy, the patient's preferred classical music (Rast or Hejaz modes) was asked by the specialist and 10 minutes of music therapy was performed according to patient's choice. Clinical data and pain scores were obtained 5, 30 and 60 minutes after music therapy. 6 sessions of music therapy were applied on different days. Patient Follow-up Form was recorded before and after each therapy. The forms were evaluated 3 times, before the application, after the 3rd and 6th application.
  Interventions: Behavioral: music therapy
- control group (No Intervention): The control group consisted of patients who only received analgesic treatment and underwent routine nursing care, and didn't have any interventions. All forms were assessed 3 times, before application, after the 3rd application and after the 6th application. The Patient Information Form and K-MASF were applied only once.

INTERVENTIONS:
Behavioral: music therapy — patients in the intervention group received music therapy in 10-minutes sessions with the support of a specialist from the Conservatory Department in the Ege University, using the Turkish classical music (Hejaz and Rast modes) accompanied by a tambour.
  Other Names: complementary therapy
  Arms: Intervention Group

SUMMARY:
Background: Palliative care services can be applied in chronic, life-threatening conditions such as cancer, and provide physical, mental and psychological support to patients worldwide. Purpose: This study aimed to investigate the effect of music on pain, anxiety, comfort and functional capacity of cancer patients received care in a palliative care unit.

Methods: The population of this randomized controlled trial consisted of cancer patients hospitalized in the Palliative Care Service of a Training and Research Hospital between July 2018-July 2019. The sample of the study included 60 patients (30 interventions/30 controls) who met the inclusion criteria. The patients in the intervention group were given a total of six music sessions, ten minutes each with the Turkish classical music in maqams (modes) of their choice (Hejaz or Rast accompanied by an expert tambour (drum) player).

DETAILED DESCRIPTION:
The incidence of chronic diseases and conditions including cancer that require a long-term treatment process and also affect the individual psychological status and quality of life has increased with a high financial burden as a result of relatively prolonged human life under the influence of contemporary medicine. Palliative care services can be applied in chronic, life-threatening conditions such as cancer, and provide physical, mental and psychological support to patients worldwide. Symptoms including pain, constipation, diarrhea, anorexia, dysphagia, nausea and vomiting, dehydration, depression, delirium, and fatigue may demonstrate in cancer patients receiving palliative care, while most of the them have complain of pain. Studies have reported that 30% of cancer patients experienced pain at the diagnosis, 50-70% of them in during treatment period, and 60-80% of them in the terminal period. It was determined in another study that 90% of patients had pain when they were hospitalized in palliative care service, and more than half of them defined the pain severity at 5 and above.

Pharmacological agents were used to manage pain control, as they had rapid effect and were easily applicable. In addition to pharmacological agents, the application of non-pharmacological interventions is important for improving the quality of life and patient comfort and reducing the symptom burden in relieving pain caused by the side effects and methods of treatment in the palliative care cancer patients. Since non-pharmacological methods could reduce pain by applying alone or in combination with drugs, the frequency of use has increased in recent years. Music therapy was used as a non-pharmacological method in many health problems as a traditional treatment and psychosocial interventions. The study was aimed to investigate the effects of music therapy on pain in patients with cancer hospitalized palliative care service. In the current study we tested the hypothesis that palliative care patients' pain management. 1. reduce the rate of pain score. 2. reduce the rate of anxiety scoe. 3. To increase the rate of comfort level. 4. To increase the rate of functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were older than 18 years old, speaking and understanding Turkish language, volunteering to participate in the study, diagnosed with cancer and hospitalized in a palliative care service, defined "moderate" or "severe" pain (>3 Visual Analog Scale scores) despite using opioid or analgesic, not in the terminal period, and not in bedridden status were included the study. Also, patients without cognitive impairment or brain metastases, and without clinical diagnosis or findings of dementia, hearing problems, agitation or delirium were enrolled the study.

Exclusion Criteria:

* Patients who were younger than 18 years old, not know speaking and understanding Turkish language, not to be volunteering to participate in the study, not diagnosed with cancer and not hospitalized in a palliative care service, Visual Analog Scale scores lower than 3 point, in the terminal period, and in bedridden status and patients with cognitive impairment or brain metastases, and with clinical diagnosis or findings of dementia, hearing problems, agitation or delirium weren't included the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
primary Outcome Measure | 3 weeks
  Patient Information Form involved questions including patients' socio-demographic data.
  Patient Follow-Up Form was for recording of vital signs and pain levels before and after the application.
  K-MASF consisted of three parts: the nature of the pain, its severity, and general pain intensity.
  GCS consisted of three levels and four dimensions. STAI was a self-assessment questionnaire consisting of short expressions. The questionnaire required patients to describe how they feel under certain conditions and to answer the scale with their feelings about these conditions.
  KPC was prognostic indicator for the patient's normal activities and functional capacity.
  There was a significant difference between the mean total pain scores, anxiety, comfort and functional capacityof the patients in the intervention and control groups before and after music therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Gönül Düzgün, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code